CLINICAL TRIAL: NCT03411707
Title: A Multicenter Clinical Trial for the Comparison Among Fecal Immunochemical Test, Stool DNA Test and Blood mRNA Test in Chinese Colorectal Cancer Screening
Brief Title: Multiple Screening Methods for the Detection of Chinese Colorectal Advanced Adenomatous Polyps and Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Changhai Hospital (Other); Tianjin Nankai Hospital (Other)
Responsible Party: Principal Investigator, Hongzhi Zou, Principal investigator, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: SC2017
Record Dates: First submitted 2018-01-20; First posted 2018-01-26 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Colorectal Cancer; Colorectal Adenomatous Polyp
Keywords: Colorectal cancer screening; Stool DNA test; Blood mRNA test
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mutiple screening test group
  Interventions: Diagnostic Test: Stool DNA test

INTERVENTIONS:
Diagnostic Test: Stool DNA test — Stool DNA test could detect specific gene methylation in stool DNA. Blood mRNA test could detect specific set of gene expression in blood.
  Other Names: Blood mRNA test; FIT Assay

SUMMARY:
The primary objective is to determine the sensitivity and specificity of two Colorectal Cancer (CRC) screening methods, including stool DNA test and blood mRNA test, for colorectal cancer in Chinese population, with colonoscopy as reference method. Lesions will be confirmed as malignant or precancerous by colonoscopy and histopathologic examination.

The secondary objective is to compare the performance of these two CRC screening methods to a commercially available FIT assay, both with respect to cancer and advanced adenoma. Lesions will be confirmed as malignant or precancerous by colonoscopy and histopathologic examination.

DETAILED DESCRIPTION:
Participants who are at high risk of developing colorectal cancer will be asked to collect two stool samples one for the stool DNA test and the other for the commercially available FIT assay, and a single blood sample for the blood mRNA test. Subjects will undergo colonoscopy within 6 months of enrollment. Representative histopathology slides from tissue biopsied or excised during colonoscopy and those from subsequent definitive surgery may be retrieved in order to be evaluated by pathologists to confirm the diagnosis and staging.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects received screening questionnaire and had been defined as high risk.
2. Subjects haven't received any treatment under colonoscopy within 10 years.

Exclusion Criteria:

1. Subjects are under the usage of specific drugs which might affect the screening test.
2. Subjects had the contraindication for colonoscopy.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants at high risk of developing colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2018-03-19 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of Multiple Screening Methods With Comparison to Colonoscopy, Both With Respect to Cancer. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhi Zou, MD, PhD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yet-sen University
Locations (3):
- China (3):
  - The Sixth Affiliated Hospital, Sun Yet-sen University, Guangzhou
  - Changhai Hospital, Shanghai
  - Tianjin Nankai Hospital, Tianjin